CLINICAL TRIAL: NCT05418361
Title: Construction of an Evidence Based Startegy for the Use of Renin Angiotensin Aldosterone System Blockers for Future Targeting of ACE2 in Treatment of COVID19
Brief Title: The Effect of RAAS Blockers on ACE2 Levels
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FAMASU/2021
Record Dates: First submitted 2022-06-10; First posted 2022-06-14 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2022-06

CONDITIONS: Renin-Angiotensin System

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ACEIs group: Patients suffer from cardiovascular diseases)controlled hypertension or heart failure ) taking ACE inhibitors
  Interventions: Drug: ACE inhibitor ,angiotensin receptor blockers
- ARBs group: Patients suffer from cardiovascular diseases)controlled hypertension or heart failure ) taking Angiotensin receptor blockers
  Interventions: Drug: ACE inhibitor ,angiotensin receptor blockers
- healthy: matched healthy controls

INTERVENTIONS:
Drug: ACE inhibitor ,angiotensin receptor blockers — patients taking ACEI or ARBs with cardiovascular disease
  Groups: ACEIs group; ARBs group

SUMMARY:
Blockage of renin-angiotensin-aldosterone system (RAAS) by angiotensin converting enzyme inhibitors (ACEI) and angiotensin receptor blockers (ARBs) is considered the first-choice of drugs for treatment of hypertension, heart failure and chronic kidney disease However, the interplay between RAAS blockers and ACE2 hasn't been fully elucidated SARS-CoV-2 is thought to infect host cells through ACE2 to cause coronavirus disease 2019 (COVID-19). Recent studies revealed that the spikes of COVID-19 could bind to the surface receptors of sensitive cells after contacting the airway surface, which may mediate virus entry into target cells and viral replication, and ACE2 might be a mediator of infection (South, Brady et al. 2020). Therefore, the imbalance in the RAAS, with a shift towards ACE/Ang II and suppression of ACE2/Ang-(1-7), may be an important mediator of COVID-19. To date, conflicting evidences were reported linking the use of RAAS blockers and the susceptibility to the virus. However, others showed that treatment with an RAAS blockers may downregulate the expression of ACE2 but have no significant effect on its activity This research importantly aimed to solve this important issue by determining the exact association between ARBs and ACE inhibitor and ACE2 activity and levels on clinical and experimental prospects.

DETAILED DESCRIPTION:
Blockage of renin-angiotensin-aldosterone system (RAAS) by angiotensin converting enzyme inhibitors (ACEI) and angiotensin receptor blockers (ARBs) is considered the first-choice of drugs for treatment of hypertension, heart failure and chronic kidney disease . The classic RAAS primarily involves 2 enzymes: renin, which cleaves angiotensinogen to the inactive decapeptide angiotensin (Ang) I; and ACE that hydrolyzes Ang I to the octapeptide Ang II, the well-known vasopressor agent . In fact, the enzymatic cascade of the RAS encompasses an ACE homolog known as ACE2. Whereas, the ACE2-dependent pathways directly yield Ang (1-9) from Ang I and degrade Ang II to Ang (1-7), which is vasodilator and acts as a feedback mechanism to antagonize the vasopressor effect of Ang II. Indeed, ACE inhibitors effectively attenuate Ang II formation and augment the levels of the heptapeptide Ang (1-7) . However, the interplay between RAAS blockers and ACE2 hasn't been fully elucidated.

SARS-CoV-2 is thought to infect host cells through ACE2 to cause coronavirus disease 2019 (COVID-19). Recent studies revealed that the spikes of COVID-19 could bind to the surface receptors of sensitive cells after contacting the airway surface, which may mediate virus entry into target cells and viral replication, and ACE2 might be a mediator of infection Therefore, the imbalance in the RAAS, with a shift towards ACE/Ang II and suppression of ACE2/Ang-(1-7), may be an important mediator of COVID-19. To date, conflicting evidences were reported linking the use of RAAS blockers and the susceptibility to the virus. However, others showed that treatment with an RAAS blockers may downregulate the expression of ACE2 but have no significant effect on its activity .

Furthermore, SARS-CoV-2 infection has largely been influenced by multiorgan involvement inducing multiple comorbidities due to the wide distribution of ACE2 thought out the whole body. In addition, hypertension, cardiovascular disease, and chronic kidney disease are supposed to be potential but unconfirmed risk factors for COVID-19 in adults and children . However, the expression of ACE2 may be lower in patients with hypertension than in people with normal blood pressure . Concluding more conflicting evidences for the association of COVID-19 with RAAS inhibitors.

Given the RAAS importance to cardiovascular and kidney physiology, and the association between chronic diseases and COVID-19, could shed light on potential relationships between ACE inhibitor and ARB use and COVID-19.

Accordingly, evidences are required to solve the question of whether ARBs and ACE inhibitor have either favorable or harmful effects on the susceptibility to SARS-CoV-2 in addition to the severity and outcomes of COVID-19 infection. This research importantly aimed to solve this important issue by determining the exact association between ARBs and ACE inhibitor and ACE2 activity and levels on clinical and experimental prospects.

ELIGIBILITY:
Inclusion Criteria:

* Patients age> 18 years
* Taking ACE II inhibitors or angiotensin II blockers (according to maximum tolerated dose specified by guidelines)
* History of essential hypertension or heart failure

Exclusion Criteria:

* patients who suffer from secondary hypertension, including idiopathic hyperaldosteronism, renal artery stenosis
* Patient reported history of severe liver disease
* a history or suspicion of alcohol or drug abuse; and mental illness
* Pregnant and breast feeding

Ages: 43 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with controlled Hypertension or heart failure presenting to Cardiac Rehabilitation Units taking ACE inhibitors or AGII blockers
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Effect of RAAS blockers on ACE2 levels | at least 6 months
  ACE2 levels in cardiovascular disease patients

CONTACTS AND LOCATIONS:
Overall Officials: ebtehal el demerdash, prof, Principal Investigator — Ain Shams University
Locations (1):
- Ainshams University, Cairo, Select A State Or Province, Egypt

REFERENCES:
- [Derived] Farid Fahmy S, El Derany MO, Khorshid H, Saleh A, El-Demerdash E. Effect of renin angiotensin blockers on angiotensin converting enzyme 2 level in cardiovascular patients. BMC Pharmacol Toxicol. 2023 Apr 14;24(1):24. doi: 10.1186/s40360-023-00667-w. PMID 37060024